CLINICAL TRIAL: NCT05555433
Title: Study of the Interest of Serum Calprotectin Determination in the Diagnosis of Spondyloarthritis and to Diferenciate With Fibromyalgia
Brief Title: Calprotectine in Spondyloarthritis
Acronym: Calprotectine
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22Rhumato01
Record Dates: First submitted 2022-09-22; First posted 2022-09-26 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Spondylarthritis
MeSH Terms: conditions — Spondylarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- active spondyloarthritis: subjects with active spondyloarthritis with a BASDAI greater than 4
  Interventions: Other: NO INTERVENTION
- remission spondyloarthritis: subjects presenting with a remission spondyloarthritis defined by a BASDAI less than 4
  Interventions: Other: NO INTERVENTION
- controls without spondyloarthritis: controls without spondyloarthritis or other chronic inflammatory rheumatism and without fibromyalgia
  Interventions: Other: NO INTERVENTION
- fibromyalgia: subjects with fibromyalgia
  Interventions: Other: NO INTERVENTION

INTERVENTIONS:
Other: NO INTERVENTION — no intervention

SUMMARY:
To date, there are no biomarkers in spondyloarthritis that can differentiate between spondyloarthritis and fibromyalgia or other pathologies. Fecal calprotectin is a biomarker that is increasingly used in inflammatory diseases of the digestive tract. A growing interest in this biomarker is emerging in rheumatology, several publications have focused on its interest in rheumatoid arthritis, highlighting an association between serum calprotectin levels and disease activity. In spondyloarthritis, a few studies seem to show that it could be a marker of disease activity. Although a 2012 study found no difference in serum calprotectin levels between subjects with spondyloarthritis and controls. Still others have shown that it could be a predictive factor of radiological evolution in the same disease key. These data support, despite the questionable results of the Klingberg study, the value of this dosage in spondyloarthritis. The objective of this work is to show that this assay could be useful to differentiate spondyloarthritis from other pathologies with similar clinical presentation such as fibromyalgia. Difficulties classically encountered in common practice in rheumatology

ELIGIBILITY:
Inclusion Criteria:

Patients in the active line of the rheumatology department with one of the following criteria:

active spondyloarthritis (BASDAI >4), or spondyloarthritis in low activity (BASDAI<4), or fibromyalgia without associated inflammatory rheumatism, or healthy subjects (without inflammatory rheumatism and without fibromyalgia. Patients who have not objected to the use of their samples

Exclusion Criteria:

Minor patient Subject not affiliated to the social security system Subject deprived of liberty Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary clinic care, rheumatology patients at the CHU de NICE
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
calprotectine rate | 5 months
  blood test

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No